CLINICAL TRIAL: NCT01798667
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Therapeutic Exploratory Clinical Trial to Evaluate the Efficacy and Safety of DA-8031 After Oral Administration in Male Patients With Premature Ejaculation
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DA-8031 in Male Patients With Premature Ejaculation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA8031_PE_II
Record Dates: First submitted 2013-01-27; First posted 2013-02-26 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — DA 8031

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): PO administration
  Interventions: Drug: Placebo
- DA-8031 dose 1 (Experimental): PO administration
  Interventions: Drug: DA-8031
- DA-8031 dose 2 (Experimental): PO administration
  Interventions: Drug: DA-8031
- DA-8031 dose 3 (Experimental): PO administration
  Interventions: Drug: DA-8031

INTERVENTIONS:
Drug: DA-8031
  Arms: DA-8031 dose 1; DA-8031 dose 2; DA-8031 dose 3
Drug: Placebo — Placebo of DA-8031, undistinguishable
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of DA-8031 and to decide the optimal dose of DA-8031 in male patients with premature ejaculation after oral administration on-demand.

The investigators hypothesized that newly-developed DA-8031 would effect in delaying ejaculation in patients with premature ejaculation (PE).

Design:

Placebo-controlled, Randomized, Double-blind, Double-dummy, Parallel group, Fixed dose design

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged with premature ejaculation for more than 6 months.
* PEDT score ≥ 11

Exclusion Criteria:

* IIEF-EF domain ≤ 21
* Serum Creatinine ≥ 2.5 mg/dl
* AST, ALT > 3*Upper limit of normal
* Subjects with hypotension(SBP/DBP<90/50mmHg) or uncontrolled hypertension(SBP/DBP>180/100mmHg)
* Subjects with chronic depression, psychiatric or schizophrenia,
* Subjects with alcohol, drug or substance abuse

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
average IELT change | From 0 week(baseline) to 8 week(end of treatment)

SECONDARY OUTCOMES:
PEP, PGI | 8 weeks
  PEP(Primary ejaculation profile), PGI(Patient-reported global impression)

CONTACTS AND LOCATIONS:
Overall Officials: Sae Woong Kim, Principal Investigator — Seoul St. Mary's Hospital; Du Geon Moon, Principal Investigator — Korea University Guro Hospital; Nam-Cheol Park, Principal Investigator — Pusan National University Hospital; Jae-Seung Paick, Principal Investigator — Seoul National University Hospital; Tai-Young Ahn, Principal Investigator — Asan Medical Center; Sung Won Lee, Principal Investigator — Samsung Medical Center; Ki Hak Moon, Principal Investigator — Yeongnam University Hospital; Kwangsung Park, Principal Investigator — Chonnam National University Hospital; Jong Kwan Park, Principal Investigator — Chonbuk National University Hospital; Dae Yul Yang, Principal Investigator — Kangdong Sacred Heart Hospital
Locations (1):
- Samsung Medical Center, Seoul, South Korea